CLINICAL TRIAL: NCT04747080
Title: The Combination of High-dose Dexamethasone and Tacrolimus Versus High-dose Dexamethasone as the First-Line Treatment of Newly-diagnosed Immune Thrombocytopenia: A Randomized, Controlled, Multicenter, Open-label Trial
Brief Title: The Combination of Tacrolimus and High-dose Dexamethasone as First-line Treatment in Adult Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Hospital (Other Government); Beijing Friendship Hospital (Other); China-Japan Friendship Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Chongqing Medical University (Other); Shanxi Bethune Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice President of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITP-PKU022
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: ITP; Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Dexamethasone; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAC and HD-DXM (Experimental): Dexamethasone 40 mg per day, 4 consecutive days (the 4-day course of dexamethasone is repeated in the case of lack of response by day 14).
  Tacrolimus is given at a dose of 0.03mg/kg·d, and the dose is adjusted to maintain the trough concentration of tacrolimus at approximately 3-5 ng/mL for 12 weeks.
  Interventions: Drug: Dexamethasone; Drug: Tacrolimus
- HD-DXM (Active Comparator): Dexamethasone 40 mg per day, 4 consecutive days (the 4-day course of dexamethasone is repeated in the case of lack of response by day 14) .
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 40 mg per day, 4 consecutive days (the 4-day course of dexamethasone is repeated in the case of lack of response by day 14).
  Other Names: HD-DXM; High-dose Dexamethasone
Drug: Tacrolimus — Tacrolimus is given at a dose of 0.03mg/kg·d, and the dose is adjusted to maintain the trough concentration of tacrolimus at approximately 3-5 ng/mL for 12 weeks.
  Other Names: TAC
  Arms: TAC and HD-DXM

SUMMARY:
Randomized, open-label, multicenter study to compare the efficacy and safety of Combination of High-dose Dexamethasone and Tacrolimus versus High-dose Dexamethasone for the first-line treatment of adults with primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicenter, randomized controlled trial of 100 adults with ITP in China. Patients were randomized to tacrolimuis plus high-dose dexamethasone and high-dose dexamethasone monotherapy group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed newly-diagnosed, treatment-naive ITP;
2. Platelet counts <30×109/L ;
3. Platelet counts < 50×109/L and significant bleeding symptoms (WHO bleeding scale 2 or above);
4. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 6 months before the screening visit;
2. Received first-line and second-line ITP-specific treatments (eg, steriods, cyclophosphamide, 6-mercaptopurine, vincristine, vinblastine, etc) ;
3. Current HIV infection or hepatitis B virus or hepatitis C virus infections;
4. Active infection;
5. Maligancy;
6. Severe medical condition (lung, hepatic or renal disorder) other than chronic ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia);
7. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period; a history of clinically significant adverse reactions to previous corticosteroid therapy
8. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test;
9. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Sustained（Durable） response | 6 months
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-month follow-up.

SECONDARY OUTCOMES:
Complete response (CR) | Day 14
  Complete response (CR) was defined as platelet count more than 100,000 per cubic millimeter and absence of bleeding.
Response (R) | Day 14
  Response (R) as platelet count more than 30,000 per cubic millimeter and at least 2-fold increase of the baseline count and absence of bleeding.
Time to response | 6 months
  The time from starting treatment to time of achievement of CR or R.
Duration of response (DOR) | 6 months
  Duration of response at 6-month follow up.
Loss of response | 6 months
  Platelet counts below 100 x 109/L or bleeding (from CR) or platelet counts below 30 x 109/L, less than 2-fold increase of baseline platelet count or bleeding (from R)
Number of participants with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale | From the start of study treatment (Day 1) up to the end of week 24.
  The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Immune Thrombocytopenia Patient Assessment Questionnaire (ITP-PAQ) | Time Frame: From the start of study treatment (Day 1) up to the end of week 24.
  In all participants ,use ITP-PAQ to assess the Health Related Quality of Life(HRQoL) before and after treatment.
Functional Assessment of Chronic Illness Therapy fatigue subscale (FACIT-F) | Time Frame: From the start of study treatment (Day 1) up to the end of week 24.
  In all participants ,use FACIT-F to assess the Health Related Quality of Life(HRQoL) before and after treatment.
Number of Participants with side effects of the drugs | Time Frame: From the start of study treatment (Day 1) up to the end of week 24.
  Side effects of the drugs included fever, headache, serum disease, infection, hypotension, rashes, infection liver injury, hypokalaemia, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided